CLINICAL TRIAL: NCT06512662
Title: Support Pathway for ENT Cancer Patients in a Support Care Day Hospital Single-centre Prospective Randomised Interventional Study
Brief Title: Support Pathway for ENT Cancer Patients in a Support Care Day Hospital
Acronym: PAKO-HDJ
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Clinique Pasteur Lanroze (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2023-18-CPL
Record Dates: First submitted 2024-07-16; First posted 2024-07-22 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-10

CONDITIONS: Otorhinolaryngologic Neoplasms
Keywords: surgery; quality of life; anxiety; supportive care
MeSH Terms: conditions — Otorhinolaryngologic Neoplasms; Anxiety Disorders | interventions — Referral and Consultation; Paramedics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (No Intervention)
- Supportive care (Experimental)
  Interventions: Procedure: Consultations with paramedics

INTERVENTIONS:
Procedure: Consultations with paramedics — Patients of experimental arm will beneficiate of supplemental consultations with paramedics intervenants at 1 month, 3 months and 6 months after surgery :
  * dietetician
  * speech therapist
  * psychologist
  * advanced practice nurse
  During these consultations, several scales will be performed to assess the patient's condition (anxiety, nutritional status, psychological condition, speech therapy status).
  Arms: Supportive care

SUMMARY:
Cancers of the upper respiratory / digestive tract are a major public health problem, ranking 5th among the most common cancers. Surgery plays a central role in the recommended treatments for this type of pathology. The surgical procedure and its after-effects can be anxiety-provoking and have a major psychological, physical and social impact on patients over the long term.

Our institution's standard protocol is based on a pre-operative supportive care day hospital. The aim of this study is to compare our current care pathway with a more extensive interdisciplinary care pathway focused on patients' needs, in order to reduce anxiety and improve the quality of life of patients undergoing surgery for cancers of the upper respiratory / digestive tract.

Our aim is to use a prospective single-centre interventional study to assess the impact of adding three post-operative day hospitals to the existing care pathway in terms of reducing anxiety and improving the quality of life of patients undergoing surgery.

ELIGIBILITY:
Inclusion Criteria:

* patient undergoing surgery for VADS cancer requiring at least one night's post-operative hospitalisation
* Understanding of spoken and written French
* Patient covered by a social security scheme

Exclusion Criteria:

* Protected patient under a protective measure or legal safeguard
* Pregnant or breast-feeding patients
* Patients suffering from major cognitive disorders
* Patients with major anxiety disorders prior to the onset of cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-10-08 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Anxiety | 1 month ; 3 months ; 6 months
  Anxiety evaluation by State Trait Anxiety Inventory (STAI) scale. It is a psychological inventory consisting of 40 self-report items on a 4-point Likert scale. The STAI measures two types of anxiety - state anxiety and trait anxiety. Higher scores are positively correlated with higher levels of anxiety.

SECONDARY OUTCOMES:
Quality of life evaluation | 1 month ; 3 months ; 6 months
  Quality of life will be evaluated by EORTC C30. The EORTC quality of life questionnaire (QLQ) is an integrated system for assessing the health-related quality of life (QoL) of cancer patients participating in international clinical trials.
pain evaluation | 1 month ; 3 months ; 6 months
  Pain will be assessed using a visual analogue scale from 0 (no pain) to 10 (worst pain imaginable).
Toxic behaviour (tobacco and alcohol) evaluation | 1 month ; 3 months ; 6 months
  Tobacco (number of cigarettes per day) and alcohol (number of units per day) consumption will be evaluated by questioning the patient.
Weight status evaluation | 1 month ; 3 months ; 6 months
  Weight statut will be determined by calculating the body mass index (BMI) and the percentage of loss weight.
nutritional status evaluation | 1 month ; 3 months ; 6 months
  Nutritional status will be evaluated using SEFI (simple evaluation of food intake) scale. This scale is a Likert scale to assess the portion eaten at mealtimes, from 0 ("I haven't eaten anything") to 10 ('I have eaten everything").
swallowing assessment | 1 month ; 3 months ; 6 months
  Swallowing is measured by Deglutition Handicap Index (DHI). It is a questionnaire with 30 questions (10 physical, 10 functional, 10 emotional) with a Likert scale from "never" to "always".
vocal status assessment | 1 month ; 3 months ; 6 months
  Vocal status is measured by Vocal Handicap Index (VHI). It is a questionnaire with 30 questions with a Likert scale from "never" to "always".

CONTACTS AND LOCATIONS:
Locations (1):
- Clinique Pasteur Lanroze, Brest, France

IPD SHARING:
Plan to Share IPD: No